CLINICAL TRIAL: NCT03419559
Title: A Phase 2 Study to Assess the Efficacy and Safety of Autologous Tumor Infiltrating Lymphocytes (LN-145) In Combination With Anti-PD-L1 Inhibitor Durvalumab (MEDI4736) in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of Autologous Tumor Infiltrating Lymphocytes (LN-145) In Combo With Durvalumab in Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The treatment landscape for NSCLC has evolved in the past year. An additional NSCLC arm will be added to the IOV-COM-202 study using TIL + pembrolizumab.
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOV-LUN-201
Record Dates: First submitted 2018-01-14; First posted 2018-02-05 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: LN-145; Cell Therapy; Autologous Adoptive Cell Transfer; Cellular Immuno-therapy; TIL; IL-2; Durvalumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Toll-Like Receptor 1; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LN-145 in combination with durvalumab (Experimental): After nonmyeloablative (NMA) lymphodepletion, patients are infused with their autologous TIL (LN-145) followed by IL-2 administration.
  Interventions: Biological: LN-145; Drug: Durvalumab

INTERVENTIONS:
Biological: LN-145 — adoptive cell therapy (ACT) with autologous TIL therapy
  Other Names: TIL, autologous tumor infiltrating lymphocytes
Drug: Durvalumab — PD-L1 antagonist monoclonal antibody
  Other Names: MEDI4736

SUMMARY:
This study is a Phase 2, open-label, multicenter study evaluating adoptive cell therapy (ACT) with autologous TIL therapy (LN-145) in combination with Anti-PD-L1 inhibitor durvalumab.

DETAILED DESCRIPTION:
LN-145 is an adoptive cell transfer therapy that utilizes an autologous TIL manufacturing process, as originally developed by the NCI. The cell transfer therapy used in this study involves patients receiving a nonmyeloablative (NMA) lymphocyte depleting preparative regimen, followed by infusion of autologous TIL followed by the administration of a regimen of IL-2.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Stage III or Stage IV NSCLC and progressed after ≤ 3 lines of prior systemic therapy in the locally advanced or metastatic setting
* Have at least 1 lesion resectable for TIL generation
* Measurable disease as defined by RECIST v1.1
* Male or female, ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and estimated life expectancy of ≥ 3 months
* Adequate bone marrow function at screening
* Adequate organ function at screening
* A washout period from prior anticancer therapy(ies) of a minimum duration is required prior to first study treatment
* Recovered from all prior anticancer therapy-related AEs to Grade 1 or less (per CTCAE v4.03) prior to enrollment
* Female patients of childbearing potential and male patients with partners of childbearing potential patient must agree to use contraception while on study and during the timeframes as specified following the last dose of study drug(s) received, or until the first dose of the subsequent anticancer therapy, whichever is longer
* Evidence of postmenopausal status or negative urine or serum pregnancy test for female premenopausal patients

Exclusion Criteria:

* History of other malignancies, except for the following: adequately treated nonmelanoma skin cancer, curatively treated in-situ cancer of the cervix, curatively-treated thyroid cancer, or other solid tumors curatively treated with no evidence of disease for ≥ 3 years
* Patients who have received prior cell therapy
* Patients who have received prior checkpoint inhibitors: such as anti-PD-1, anti-PD-L1 inhibitors, and durvalumab
* Active or prior documented autoimmune or inflammatory disorders
* History of primary or acquired immunodeficiency syndrome, history of allogeneic organ transplant that requires therapeutic immunosuppression
* Received live or attenuated vaccination within 28 days prior to the start of NMA-LD
* Patients with a history of hypersensitivity to any component of the study drugs
* Mean QT interval ≥ 470 msec
* Patients who have a left ventricular ejection fraction (LVEF) of < 45% or who are New York Heart Association (NYHA) Class 2 or higher
* Serious illnesses or medical conditions, which would pose increased risk for study participation and/or compliance with the protocol
* Patients who have obstructive or restrictive pulmonary disease and have a documented FEV1 (forced expiratory volume in 1 second) of ≤ 60%
* Active central nervous system metastases and/or leptomeningeal disease
* Female patients who are pregnant or breastfeeding
* Active infection including tuberculosis (TB), hepatitis B, hepatitis C, or HIV
* Current or prior use of immunosuppressive medication within 28 days before the first dose of study treatment, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | A maximum of 24 months
  To evaluate efficacy using the objective response rate (ORR)
≥ Grade 3 Treatment-Emergent Adverse Event | A maximum of 24 months
  To evaluate the safety as measured by any ≥ Grade 3 treatment-emergent adverse event (TEAE) rate

SECONDARY OUTCOMES:
Duration of Response | A maximum of 24 months
  To further evaluate efficacy such as the duration of response (DOR)
Progression Free Survival | A maximum of 24 months
  To further evaluate efficacy such as progression free survival (PFS)
Overall Survival | A minimum of 5 years
  To further evaluate efficacy such as overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Iovance Medical Monitor, Study Director — Iovance Biotherapeutics, Inc.
Locations (8):
- United States (8):
  - University of California San Diego, Moores Cancer Center, La Jolla, California
  - University of California, Los Angeles, Santa Monica Hematology/Oncology, Los Angeles, California
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Karmanos Cancer Institute, Detroit, Michigan
  - Morristown Medical Center Atlantic Hematology Oncology, Morristown, New Jersey
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No